CLINICAL TRIAL: NCT05278520
Title: Studies on the Complex Molecular Etiology and Cellular Landscape of Hip Osteoarthritis
Brief Title: Complex Molecular Etiology and Cellular Landscape of Hip Osteoarthritis
Acronym: OASEQ
Status: Recruiting | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Turku University Hospital (Other Government); Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Lea Mikkola, Principal Investigator, University of Turku
Other Study IDs: 2022OASEQ
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Hip; Rheumatoid Arthritis
Keywords: Single-cell RNA sequencing; Spatial transcriptomics; Osteoarthritis; Rheumatoid arthritis; Spatial proteomics
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Hip joint synovial tissues and bone, peripheral blood mononuclear cells, serum, plasma, and whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- OA cases: Fifty adult patients who have hip osteoarthritis.
  Interventions: Procedure: Total hip arthroplasty
- RA cases: Forty adult patients who have rheumatoid arthritis in the hip joint.
  Interventions: Procedure: Total hip arthroplasty
- Non-arthritic controls: Twenty adult patients who go through trauma-based emergency total hip arthroplasty and do not have arthritis.
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — Hip joint replacement surgery. Elective for RA and OA cases.

SUMMARY:
The purpose of this study is to cast light on the highly complex etiology and cellular landscape of hip osteoarthritis by utilising single-cell and spatial omics.

DETAILED DESCRIPTION:
The specific objectives of this project are:

1. Using the latest single-cell RNA sequencing (scRNAseq) techniques the investigators aim to A) characterize what kind of cell populations are found in different synovial tissues and blood derived samples of OA patients, B) determine how the cell composition differs between arthritic and corresponding non-arthritic tissues, C) map the transcriptional and regulatory landscape of the cells mentioned in A and B focusing on the inflammatory responses, D) determine what are the key molecular pathways activated in OA.
2. To determine if some of the blood-derived immune cell populations or their products could be used as biomarkers for OA.
3. To map the whole transcriptome and proteome of OA and non-arthritic control tissue while keeping the morphological context with spatial omics technologies.
4. Further differentiation and identification of OA endotypes utilizing the single-cell and spatial omics data.

The project includes a Rheumatoid sub-study where the main objective is to compare arthritic tissue and peripheral blood constituents between OA and rheumatoid arthritis patients to explore the differences in the disease mechanisms.

ELIGIBILITY:
Inclusion Criteria for the main (OA) study:

Cases: Adult patients with osteoarthritis in the hip joint and who are going through an elective total hip arthroplasty.

Controls: Non-arthritis adult patients who are going through a trauma-based emergency total hip arthroplasty.

----

Inclusion Criteria for the Rheumatoid sub-study:

Adult patients with rheumatoid arthritis in the hip joint and who are going through an elective total hip arthroplasty.

----

Exclusion Criteria:

* The body mass index must be below 35
* Age < 18 or > 74
* The OA patients may not have diabetes, rheumatoid arthritis (RA), or metabolic syndrome.

For the Rheumatoid sub-study, the exclusion criteria are the same as above except for the RA.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients of the HUS (Joint Authority of the Helsinki and Uusimaa Hospital District) Center of Arthroplasty and the Orto Surgical Hospital of Turku University.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of cell populations in OA | Starting during the first quarter of 2025, ending by the last quarter of 2026.
  Characterization of cell populations found in different synovial tissues and blood derived samples of OA patients utilising single-cell RNA sequencing solutions.
Comparison of cell populations between OA cases and controls | Starting during the first quarter of 2025, ending by the last quarter of 2026.
  The investigators will determine how the cell composition differs between arthritic and corresponding non-arthritic tissues utilising single-cell RNA sequencing solutions.
Cellular landscape in OA | Starting during the last quarter of 2024, ending by the last quarter of 2026.
  The investigators will map the transcriptional, regulatory and protein landscape of OA at single-cell and tissue (spatial) level.
Key molecular pathways of OA | Starting during the last quarter of 2025, ending by the last quarter of 2027.
  The investigators will determine what are the key molecular pathways activated in OA.
Comparison of disease mechanisms between RA and OA | Starting during the last quarter of 2024, ending by the last quarter of 2028.
  In the Rheumatoid sub-study the investigators will explore the differences in the disease mechanisms between OA and RA by comparing synovial tissues and peripheral blood sample constituents.

SECONDARY OUTCOMES:
Biomarkers for OA | Starting during the second half of 2026, ending by the last quarter of 2028.
  The investigators will investigate if some of the blood-derived immune cell populations or their products could be used as biomarkers for OA.
OA endotypes | Starting during the first half of 2025, ending by the second half of 2027.
  The investigators aim to identify and further differentiate OA endotypes by utilizing the single-cell and spatial data.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Mikkola, PhD, Principal Investigator — Turku Bioscience, University of Turku
Locations (4):
- Finland (4):
  - PET-centre, University of Turku, Turku, Southwest Finland
  - Turku Bioscience, University of Turku, Turku, Southwest Finland
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital, Espoo, Uusimaa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rydgren E, Kotilainen SK, Piipponen M, Lönnberg T, Mikkola L. COMPARISON OF TWO HIGH-RESOLUTION SPATIAL TRANSCRIPTOMICS TECHNOLOGIES TO STUDY SYNOVIAL IMMUNE INFILTRATION IN OSTEOARTHRITIS AND RHEUMATOID ARTHRITIS Osteoarthritis and Cartilage, Volume 33, Issue 6, 2025, page 816. https://doi.org/10.1016/j.joca.2025.03.079